CLINICAL TRIAL: NCT04273022
Title: The Effect of Exercise on Resting Biomarkers in Subjects With Sickle Cell Trait
Brief Title: Effect of Exercise on Biomarkers in SCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Collaborators: American Society for Clinical Laboratory Science (Unknown)
Responsible Party: Principal Investigator, Tim Randolph, PhD, MT (ASCP), Professor, St. Louis University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 30577
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Sickle Cell Trait
Keywords: Sickle Cell Trait
MeSH Terms: conditions — Sickle Cell Trait | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: SCT subjects will be evaluated for activation of five physiological pathways by measuring 15 biomarkers before and after a single bout of moderate exercise. The control group will confirm normal biomarkers at rest and determine the natural response to moderate exercise.
Who Masked: Outcomes Assessor
Masking Description: Blood and urine samples will be assigned a random code. Testing personnel will be blinded to whether samples are pre- or post-exercise and whether from the SCT or control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCT Group (Experimental): Fifteen SCT subjects will be recruited, consented, screened, and enrolled if they meet inclusion and exclusion criteria. Each subject will undergo a single bout of standardized exercise on a treadmill. Subjects will self-select treadmill speed at 0% grade and begin. After 3 minutes the grade will be increased by 1% every 2 minutes until the target heart rate (70% of heart rate reserve) is reached. Speed and grade will be held constant for 15 minutes, marking the end of the session.
  Interventions: Other: Exercise
- Control Group (Active Comparator): Five healthy subjects will be recruited, consented, screened, and enrolled if they meet inclusion and exclusion criteria. Each subject will undergo a single bout of standardized exercise on a treadmill. Subjects will self-select treadmill speed at 0% grade and begin. After 3 minutes the grade will be increased by 1% every 2 minutes until the target heart rate (70% of heart rate reserve) is reached. Speed and grade will be held constant for 15 minutes, marking the end of the session.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — A single bout of standardized, moderate exercise

SUMMARY:
This study measures the effect of exercise on a variety of biomarkers in blood and urine selected to evaluate the physiological pathways of hemolysis, myolysis, thrombosis, inflammation, and renal function in subjects with sickle cell trait. These pathways have been shown to be associated with adverse events in athletes and warfighters with SCT upon protracted, repeated, strenuous exertion. Changes in biomarkers post-exercise compared to pre-exercise (and compared to healthy controls) suggest activation of the associated pathway(s) which may contribute to exercise-related events in athletes and warfighters and subclinical complications in non-athletes.

DETAILED DESCRIPTION:
Subjects with sickle cell trait and healthy controls will be subjected to a single bout of moderate, controlled exercise on a treadmill. Blood and urine samples will be collected before exercise, immediately after exercise, and 24 hours after exercise. Fifteen biomarkers, three selected to evaluate each of the five physiologic pathways previously listed, will be tested at each of the three time points. Abnormal biomarkers before exercise suggest chronic pathway activation while exacerbated levels after exercise suggest further activation stimulated by exercise. Biomarker levels 24 hours post-exercise will be used to evaluate continued pathway activation or pathway recovery. By definition, 95% of health controls will show normal biomarker levels pre-exercise and biomarker patterns post-exercise will serve as the expected standard by which to compare the test subjects.

ELIGIBILITY:
Inclusion Criteria: Sickle Cell Trait Group (AS)

* Health subjects with sickle cell trait (AS)
* Ages 18-70 years

Inclusion Criteria: Control group (AA)

* Healthy subjects without sickle cell trait (AA)
* Ages 18-70 years

Exclusion Criteria: Sickle Cell Trait group (AS) AND healthy controls (AA).

Subjects will be excluded if they:

* weigh less than 110 pounds,
* are pregnant,
* have hemoglobinopathies (other than sickle cell trait) as determined by Hb electrophoresis,
* have other self-reported conditions known to cause blood coagulation activation, myocyte destruction, hemolysis, chronic inflammation, or renal disease
* any condition that places subjects at risk during exercise.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in reticulocyte count | Immediately before, immediately after, & 24 hours after a single bout of submaximal exercise on a treadmill
  Reticulocytes will be counting using a manual microscopic method (New Methylene Blue) from blood collected in EDTA and reported as percentage of reticulocytes per 100 erythrocytes. Elevated reticulocytes suggest the bone marrow response to hemolysis.
Change in erythrocyte morphology amounts | Immediately before, immediately after, & 24 hours after a single bout of submaximal exercise on a treadmill
  Blood collected in EDTA will be smeared on a microscope slide, stained with Wright stain, and analyzed for abnormal morphologic forms with a particular interest in sickle cells. Each abnormal erythrocyte morphologic form will be reported on a Likert scale from 1-4+ as follows: 1+ (few abnormal cells); 2+ (approximately 1/3 abnormal cells); 3+ (approximately 1/2 abnormal cells); 4+ (>1/2 abnormal cells). Increasing numbers of sickle cells in response to exercise may be associated with increased hemolysis, myocyte destruction, inflammation, initiation of coagulation, and renal dysfunction.
Change in haptoglobin level | Immediately before, immediately after, & 24 hours after a single bout of submaximal exercise on a treadmill
  Haptoglobin will be measured on serum collected in a clot tube and reported as mg/dL (milligrams/deciliter) using a radial immunodiffusion method. Low haptoglobin levels suggest intravascular hemolysis.
Change in potassium (K+) level | Immediately before, immediately after, & 24 hours after a single bout of submaximal exercise on a treadmill
  Potassium will be measured in serum collected in a clot tube, analyzed by ion selective electrode, and reported in mEq/L (milliequivalents/liter) or mmole/L (millimoles/liter). Elevated potassium levels suggest intravascular hemolysis.
Change in creatine kinase (CK) level | Immediately before, immediately after, & 24 hours after a single bout of submaximal exercise on a treadmill
  Creatine kinase will be measured in serum from a clot tube, analyzed spectrophotometrically by enzyme kinetics and reported in U/L (units [of enzyme activity]/liter. Elevated creating kinase levels suggest myocyte destruction in the post-exercise environment.
Change in serum myoglobin level | Immediately before, immediately after, & 24 hours after a single bout of submaximal exercise on a treadmill
  Myoglobin will be measured in urine, analyzed by electrochemiluminescent Immunoassay or nephelometry and reported in ng/mL (nanograms/milliliter). Elevated myoglobin suggests myocyte destruction.
Change in urine myoglobin level | Immediately before, immediately after, & 24 hours after a single bout of submaximal exercise on a treadmill
  Myoglobin will be measured in urine, analyzed by electrochemiluminescent immunoassay or nephelometry and reported in mg/L (milligrams/liter). Elevated myoglobin suggests myocyte destruction.
Change in D-dimer level | Immediately before, immediately after, & 24 hours after a single bout of submaximal exercise on a treadmill
  D-dimer will be measured in citrated plasma, analyzed by immunoturbidimetry and reported in ug/mL (micrograms/milliliter). Elevated D-dimer suggests the initiation of abnormal clotting or an inflammatory reaction.
Change in fibrin monomer level | Immediately before, immediately after, & 24 hours after a single bout of submaximal exercise on a treadmill
  Fibrin monomer will be measured in citrated plasma, analyzed by the hemeagglutination method, and reported as negative (normal) or positive (abnormal). Elevated fibrin monomers suggest the initiation of coagulation.
Change in antithrombin III (ATIII) level | Immediately before, immediately after, & 24 hours after a single bout of submaximal exercise on a treadmill
  Antithrombin III will be measured in serum from a clot tube, analyzed by radial immunodiffusion, and reported in mg/dL (milligrams/deciliter). Low antithrombin III levels suggest the initiation of coagulation.
Change in C-reactive protein (CRP) level | Immediately before, immediately after, & 24 hours after a single bout of submaximal exercise on a treadmill
  C-reactive protein will be measured in serum from a clot tube, analyzed by radial immunodiffusion, and reported in mg/dL (milligrams/deciliter). Elevated C-reactive protein suggest an inflammatory reaction.
Change in erythrocyte sedimentation rate (ESR) level | Immediately before, immediately after, & 24 hours after a single bout of submaximal exercise on a treadmill
  Erythrocyte sedimentation rate will be measured on whole blood collected in EDTA using the Wintrobe method and reported in mm/hr (millimeters/hour). An elevated erythrocyte sedimentation rate suggests an inflammatory reaction.
Change in 11-dehydrothrombaxaneB2 (11-DTXB2) level | Immediately before, immediately after, & 24 hours after a single bout of submaximal exercise on a treadmill
  11-dehydrothromboxane B2 will be measured in urine using an enzyme-linked immunosorbant assay (ELISA) and will be reported as pg/mL of creatinine (picogram/milliliter of creatinine). 11-dehydrothrombozane B2 is a direct measure of platelet activation and an indirect measure of an inflammatory reaction.
Change in complete urinalysis results | Immediately before, immediately after, & 24 hours after a single bout of submaximal exercise on a treadmill
  A 10 parameter dipstick and a microscopic examination of urine will be performed on each urine sample collected. Each of the 10 dipstick parameters will be reported according to the package insert. We will pay particular attention to intact RBCs on the dipstick and sediment as an indicator of glomerular dysfunction, free hemoglobin as an indicator of hemolysis, elevated protein as an indicator of renal dysfunction or hemoglobinuria or myoglobinuria (hemolysis), and specific gravity interpreted in the context of blood and protein levels (and glucose) as an indicator of renal dysfunction.
Change in microalbumin level | Immediately before, immediately after, & 24 hours after a single bout of submaximal exercise on a treadmill
  Microalbumin will be measured in urine with a dipstick using the sulfonephthalein dye method as an indicator of renal dysfunction and reported in mg/L (millighrams/liter).

CONTACTS AND LOCATIONS:
Overall Officials: Tim R Randolph, PhD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
A final de-identified database of study data will be generated and used for data sharing. Written data sharing requests from outside researchers will be reviewed by the PI and other members of the research team. Sharing will require a written agreement between the involved parties, which specifies the following: (1) what data will be shared, (2) who will have access to the shared data, (3) how the data will be shared and where the shared data will be stored (including details about security for data transfer and storage), (4) when the data will be shared, and (5) details about the data (i.e. data formats/transformations for sharing, meta-data to be included, etc.). The agreement will also require a commitment to using the data only for the specified research purposes and a commitment to destroying or returning the data after analyses are completed. Before sharing occurs, the written agreement will also be reviewed and approved by the the appropriate University units.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available beginning 3 months after article publication for a period of 3 years after article publication
Access Criteria: Proposals from outside investigators requesting permission to access data can be made to the PI at tim.randolph@health.slu.edu